CLINICAL TRIAL: NCT00558922
Title: A Phase 1-2, Multicenter, Open-Label Study of the X-Linked Inhibitor of Apoptosis (XIAP) Antisense AEG35156 Given in Combination With Carboplatin and Paclitaxel in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: A Phase 1-2 XIAP Antisense AEG35156 With Carboplatin and Paclitaxel in Patients With Advanced Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Unacceptable Neurotoxicity (2 cases)
Sponsor: Aegera Therapeutics (Industry)
Responsible Party: Jacques Jolivet, MD, Senior VP Clinical, Aegera Therapeutics Inc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AEG35156-203
Record Dates: First submitted 2007-11-13; First posted 2007-11-15 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Lung; Non small cell; antisense; oligonucleotide; paclitaxel; carboplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — AEG 35156

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AEG35156 — AEG35156 will be given as a 2-hour intravenous infusion once weekly with a 2-hour loading dose given daily in the 2 days immediately prior to Day 1 (on Days -2 and -1) only in Cycle 1.

SUMMARY:
This is an open-label multicenter, phase 1-2 study. Following determination of the recommended AEG35156 dose in combination with carboplatin and paclitaxel in the initial Phase 1 part of this study, additional patients will be enrolled in the Phase 2 part of the study to assess the activity of the combination in advanced non small cell lung cancer.

DETAILED DESCRIPTION:
Apoptotic induction in cancer cells is a sought after therapeutic goal. Most successful anticancer agents activate apoptosis pathways in the cancers they treat. Apoptotic pathways in cells appear to converge on a single family of enzymes, the caspases, which are proteases that dismantle the cell in an orderly, non-inflammatory fashion, resulting in cell death. The X-linked Inhibitor of Apoptosis (XIAP) is the only known cellular inhibitor of caspases, its over expression thereby blocking the principal means of apoptosis. A wide range of evidence indicates that cellular overexpression of members of the IAP family is a fundamental means by which many cancer cells evade death, even in the presence of strong extrinsic (death receptor-mediated) and intrinsic (mitochondria-mediated) apoptotic cues. The inhibition of cellular XIAP activity, specifically in cancer cells under stress and primed for apoptosis by chemotherapeutic agents, is viewed as a powerful means of tipping the balance towards cell death. In particular, XIAP down regulation has been shown to enhance taxane cytotoxicity preclinically. AEG35156 is a second generation antisense which targets XIAP mRNA to lower XIAP levels and the apoptotic threshold of cancer cells, enhancing their sensitivity to intrinsic death and chemotherapy. AEG35156 may thus enhance the anticancer activity of carboplatin and paclitaxel in patients with advanced non small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed stage IIIB (malignant pleural effusion) or stage IV non small cell lung cancer who are candidates for carboplatin and paclitaxel chemotherapy for metastatic disease
* ECOG performance < 2
* One or more tumors measurable by RECIST criteria on CT scan or MRI (Phase 2 part only)
* Life expectancy of at least 3 months
* Age > 18 years
* Signed, written IRB-approved informed consent
* A negative serum pregnancy test (if applicable)
* Acceptable liver function:
* Bilirubin within normal limit
* AST (SGOT), ALT (SGPT) and Alkaline phosphatase < 2.0 times the institution's upper limit of normal
* Acceptable renal function:
* Serum creatinine within normal limits, OR calculated creatinine clearance > 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Acceptable hematologic status:
* Granulocyte > 1500 cells/uL
* Platelet count > 100,000 plt/uL
* Hemoglobin > 9.0 g/dL
* Acceptable coagulation status:
* PT within normal limits
* PTT within normal limits
* For women of child-bearing potential, the use of effective contraceptive methods during the study
* Prior radiotherapy is allowed provided disease progression outside the radiation field has been documented, treatment completed at least 2 weeks prior to registration and less than 25% of the bone marrow exposed

Exclusion Criteria:

* Prior chemotherapy for metastatic disease.
* Patients with prior history of peripheral neuropathy
* Patients with hypersensitivity to platinum containing compounds, mannitol or drugs formulated in Chremophor EL.
* Active progressive brain metastases including the presence of any related symptoms or need for corticosteroids. A CT or MRI scan of the head is necessary in patients with a history of brain metastases to document the stability of prior lesions.
* Known bleeding diathesis
* Pregnant or nursing women. NOTE: Women of child-bearing potential must agree to use adequate contraception (sterile or surgically sterile; hormonal or barrier method of birth control; or abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Men who are unwilling to use acceptable forms of birth control when engaging in sexual contact with women of child bearing potential
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* Known infection with HIV, hepatitis B, or hepatitis C
* Serious nonmalignant disease that could compromise protocol objectives in the opinion of the investigator and/or the sponsor
* Patients who have received any other investigational agent within the last 30 days. Subjects who have used a previous antisense oligonucleotide in the last 90 days will be excluded
* Unwillingness or inability to comply with procedures required in this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-09; Primary Completion 2009-08 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
To determine the recommended dose of AEG35156 when used in combination with carboplatin and paclitaxel and if the dose can enhance the response rate of carboplatin and paclitaxel in patients with advanced non small cell lung cancer. | 2 years

SECONDARY OUTCOMES:
To determine progression-free survival. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Jotte, MD, Principal Investigator — Rocky Mountain Cancer Centers; Jacques Jolivet, MD, FACP, Study Director — Aegera Therapeutics, Inc.
Locations (6):
- United States (6):
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Central Indiana Cancer Center, Indianapolis, Indiana
  - Dayton Oncology & Hematology, P.A., Dayton, Ohio
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Virginia Oncology Associates, Norfolk, Virginia
  - Northwest Cancer Specialists, P. C., Vancouver, Washington